CLINICAL TRIAL: NCT01130428
Title: Pilot Study on the Effect of Mechanical Stimulation of Bone on ATP Release in Humans in Vivo
Brief Title: Mechanical Bone Stimulation and Adenosine 5'-Triphosphate (ATP) Release in Humans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Research Center for Ageing and Osteoporosis, Copenhagen University Hospital, Copenhagen, Denmark. (Unknown); University of Sheffield (Other)
Responsible Party: PC Dagnelie PhD, Maastricht University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MEC 10-3-026; ATPBone-WP7.2
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Osteoporosis
Keywords: Mechanical stimulation; Vibration platform; Bone metabolism; ATP release
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): As a mechanical intervention, we will use a vibration platform to administer mechanical stimulation to the forearm of subjects (see Figure 1). All subjects will participate in a single experiment during which they will receive the mechanical intervention a fixed dose of; the duration of an experiment is approximately three hours.
  Interventions: Device: Juvent 1000 Vibration Platform

INTERVENTIONS:
Device: Juvent 1000 Vibration Platform — As a mechanical intervention, mechanical stimulation in the form of vibration will be administered to the forearm using a Juvent 1000 Vibration Platform (Juvent Medical, Inc., Lakeland, FL, USA), which is a non-medicinal product. The device produces gentle, low-magnitude mechanical signals in the form of low-amplitude vertical displacements at a high frequency.
  The intervention in the present study will be given at a fixed dosage that is defined by the intensity of vibration: frequency: 90 Hz, amplitude: 10 µm (~3.0 g). The mechanical stimulation will be administered in an intermittent fashion, as it has been shown that inserting short rest periods between loading cycles enhances the efficacy of mechanical loading [38]. Thus, the mechanical stimulation will be administered for three times 10 minutes (i.e. the vibration platform turned on), with 10-minute rest periods in between (i.e. the vibration platform turned off); the intervention will have a total duration of 50 minutes.

SUMMARY:
Rationale: Mechanical loading is well-known to have a strong anabolic effect on bone. It has therefore been proposed that a mechanical intervention could be an effective non-pharmacological approach to treat bone loss associated with conditions such as osteopenia and osteoporosis. Data from in vitro experiments indicate that the purine nucleotide adenosine 5'-triphosphate (ATP) is released by bone cells and mediates cellular crosstalk via P2 purinergic receptors in response to mechanical stimulation. ATP release by bone cells may thus be part of a general mechanism by which mechanical loading ultimately results in increased bone formation, but this remains to be investigated in humans in vivo. The investigators hypothesize that a mechanical intervention in humans leads to a rise in systemic ATP concentrations due to ATP release from bone.

Objective: To investigate in vivo whether a measurable increase in systemic ATP levels occurs in response to mechanical stimulation of bone in humans.

Study design: Intervention study with a non-randomized, non-blinded design. All subjects will participate in a single experiment, lasting approximately 3 hours, during which the subjects will receive a mechanical intervention at a fixed dose.

Study population: Maximally 10 healthy human volunteers (18-35 y). Intervention: Subjects will receive a gentle and safe mechanical intervention, which will be administered by means of a Juvent 1000 Vibration Platform delivering low-magnitude mechanical stimuli (i.e. vibrations) to the forearm. The mechanical stimulation will be administered at a frequency of 90 Hz and amplitude of 10 µm in an intermittent fashion, i.e. three 10-minute periods of stimulation with 10-minute rest periods in between.

Main outcome parameters: As the primary outcome parameter, a change in extracellular ATP concentrations as a result of the mechanical intervention will be assessed systemically.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human volunteers;
* Age 18-35 years;
* Cannulation of veins in forearm possible;
* Written informed consent.

Exclusion Criteria:

* Metabolic bone disease (osteoporosis, Paget's Disease, hyperparathyroidism, osteomalacia) or any other condition affecting bone metabolism (e.g. corticoid-treated rheumatoid arthritis);
* Recent bone fracture of any kind ≤ 12 months preceding the study;
* Blood donors.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in systemic ATP levels in response to mechanical stimulation | Pre-post treatment comparison
  As the primary outcome parameter, ATP release from bone after a mechanical intervention will be investigated in humans in vivo by assessing a change in systemic concentrations of ATP and its metabolites in response to mechanical stimulation as an objective outcome measure. A change in levels of ATP (or its metabolites) is defined as the average of three concentrations after the intervention minus the average of three concentrations before the intervention (i.e. baseline).

CONTACTS AND LOCATIONS:
Overall Officials: PC Dagnelie, PhD, Study Chair — Maastricht University Medical Center, Department of Epidemiology; MJL Bours, PhD, Principal Investigator — Maastricht University Medical Center, Department of Epidemiology
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- See also: website EU project on the role of purinergic P2 receptor signalling in bone metabolism and osteoporosis — http://www.atpbone.org/